CLINICAL TRIAL: NCT02106247
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of BI 1181181 in Young Healthy Male Volunteers (Randomised, Double-blind, Placebo-controlled Within Dose Groups Phase I Trial)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Oral Doses of BI 1181181 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1344.20; 2013-004563-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (3):
- 1 BI 1181181 low dose (Experimental): tablet
  Interventions: Drug: BI 1181181 low dose
- BI 1181181 high dose (Experimental): tablet
  Interventions: Drug: BI 1181181 high dose
- Placebo (Experimental): tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1181181 high dose — two tablet
  Arms: BI 1181181 high dose
Drug: BI 1181181 low dose — one tablet
  Arms: 1 BI 1181181 low dose
Drug: Placebo — tablet
  Arms: Placebo

SUMMARY:
To assess the reduction of ß-amyloid levels in cerebrospinal fluid and plasma and to evaluate pharmacokinetics, safety and tolerability following single oral doses of BI 1181181.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator´s assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age 18 to 50 years (incl.)
3. BMI 18.5 to 29.9 kg/m2 (incl.)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure < 90 mmHg and >= 140 mmHg at screening in supine position
3. Repeated measurement of diastolic blood pressure < 55 and >= 90 mmHg at screening in supine position
4. Repeated measurement of pulse rate < 40 bpm and > 90 bpm at screening
5. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
6. Any evidence of a concomitant disease judged clinically relevant by the investigator
7. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
8. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial drug
9. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
10. History of relevant orthostatic hypotension, fainting spells, or blackouts
11. Chronic or relevant acute infections
12. Positive testing on infectious diseases
13. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)
14. Intake of drugs with a long half-life (>24 hours) within 30 days or less than 10 halflives of the respective drug prior to administration of trial medication
15. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial
16. Participation in another trial with investigational drug administration within 60 days prior to administration of trial medication
17. Smoker (more than 10 cigarettes or 3 cigars or 3 pipes/day)
18. Inability to refrain from smoking on trial days
19. Alcohol abuse (consumption of more than 40 g per day)
20. Drug abuse
21. Positive testing in the alcohol breath test or the drug screening test
22. Blood donation (more than 100 mL within 30 days prior to administration of trial medication or during the trial)
23. Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
24. Inability to comply with dietary regimen of trial site
25. At screening, a marked baseline prolongation of QT/QTc interval (such as repeated demonstration of a QTcF interval >450 ms) or any other relevant ECG finding
26. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
27. Abnormal parameters for thyroid hormones (T3, T4, TSH), coagulation parameters (partial thromboplastin time (aPTT), prothrombin time (PT) and fibrinogen (retests prior inclusion are allowed))
28. Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
29. Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two month after the trial completion. Acceptable methods of contraception comprise barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive for at least two month prior trial participation)
30. History of retinopathy
31. Any history or present disease of the central nervous system, the spinal cord or the spinal column, which could provoke complications with procedure of the lumbar catheterization/intrathecal punction
32. Signs of intracranial overpressure as determined by funduscopy

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
%-change from baseline of Aß1-40 in cerebrospinal fluid at the end of the dosing interval (i.e., 24 hrs post dose) (PoM) | up to 24 h

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma and cerebrospinal fluid over the time interval from 0 to the last quantifiable data point) | up to 72 h
Cmax (maximum measured concentration of the analyte in plasma and cerebrospinal fluid) | up to 72 h
AUC0-infinity (area under the concentration-time curve of the analyte in plasma and cerebrospinal fluid (if possible) over the time interval from 0 extrapolated to infinity) | up to 72 h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1344.20.32001 Boehringer Ingelheim Investigational Site, Antwerp, Belgium